CLINICAL TRIAL: NCT06793488
Title: Neural Mechanisms of Anxiety During Early and Protracted Abstinence in Alcohol Use Disorder
Brief Title: Anxiety During Abstinence in AUD
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, A. Benjamin Srivastava, Assistant Professor of Clinical Psychiatry, Columbia University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: AAAV4012; K23AA030355 (NIH)
Record Dates: First submitted 2025-01-21; First posted 2025-01-27 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Alcohol Use Disorder
Keywords: fMRI; disulfiram; withdrawal; anxiety; abstinence
MeSH Terms: conditions — Alcoholism; Anxiety Disorders | interventions — Disulfiram; Magnetic Resonance Imaging

STUDY DESIGN:
Intervention Model Description: Participants with alcohol use disorder (n=40) will be administered disulfiram for 3 months, which will serve to facilitate abstinence from alcohol in order to study the mechanisms of anxiety during early and protracted abstinence in alcohol use disorder. The will undergo fMRI scanning after 1 week and 3 months of disulfiram. Participants will be observed taking disulfiram both remotely (4/5 work days/week) and in person 1 day/week. Healthy volunteer participants (n=20) will not receive disufiram and will only be scanned once.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Participants with Alcohol Use Disorder (Experimental): Participants with Alcohol Use Disorder (AUDP) will be participants (n=40) ages 21-55 with alcohol use disorder (AUD) who are seeking treatment for AUD. They will undergo 3 months of treatment with disulfiram 250mg daily with supervised dosing and undergo fMRI scanning after 1 week and 3 months of disulfiram treatment.
  Interventions: Drug: Disulfiram 250 mg; Diagnostic Test: functional MRI
- Healthy volunteer participants (Other): Healthy volunteer participants will be participants (n=20) ages 21-55 without a history of alcohol or other substance use disorders. They will undergo fMRI scanning once.
  Interventions: Diagnostic Test: functional MRI

INTERVENTIONS:
Drug: Disulfiram 250 mg — Disulfiram will be used in Participants with Alcohol Use Disorder only to facilitate abstinence.
  Other Names: antabuse
  Arms: Participants with Alcohol Use Disorder
Diagnostic Test: functional MRI — Participants will undergo fMRI scanning. Participants with alcohol use disorder will undergo scanning after 1 week and 3 months of disulfiram maintenance. Healthy volunteer participants will undergo scanning once.
  Other Names: fMRI

SUMMARY:
The goal of this study is to better understand the underlying neurobiological basis of anxiety that emerges during abstinence in patients with alcohol use disorder (AUD). The main questions it aims to answer are:

1. To characterize anxiety itself as well as anxiety related-neurobiological circuitry in early abstinence in AUD
2. To examine how anxiety and anxiety related-neurobiological circuitry change over the course of abstinence in AUD

Researchers will recruit both participants with AUD and healthy volunteers.

The participants with AUD will be prescribed disulfiram, a medication that helps participants with AUD stay abstinent. Healthy volunteers will not receive antabuse. Patients with AUD will undergo fMRI scanning both after 1 week and 3 months of disulfiram treatment. Healthy volunteers will undergo fMRI once.

DETAILED DESCRIPTION:
This study will recruit 40 treatment-seeking participants with AUD ("AUDP") and 20 age matched healthy volunteer participants (HVP). AUDP will be initiated on disulfiram, a medication FDA approved for alcohol use disorder that is a first line treatment for maintenance of abstinence from alcohol, to facilitate and help ensure abstinence from alcohol and will undergo functional MRI scanning at two timepoints: 1) 8-14 days after the last drink ("early abstinence") and 2) after three months of abstinence ("protracted abstinence"). HVP will be scanned once. The investigators will examine the functioning of the Anterior Insula (AI), Bed Nucleus of the Stria Terminalis (BNST), and Dorsolateral Prefrontal Cortex (DLPFC) during a task that evokes anxiety while anticipating an uncertain threat ("threat-anxiety") as well as resting state functional connectivity (RSFC) between AI-BNST and AI-DLPFC to measure whether there are neuroplastic changes in these circuits that occur during abstinence. These changes in anxiety circuit activity and connectivity will be related to changes in current anxiety symptoms.

ELIGIBILITY:
Inclusion Criteria (Participants with Alcohol use Disorder):

1. Between the ages of 21 and 55
2. Right-handed
3. Able to perform informed consent and comply with study
4. Seeking treatment for AUD
5. Meets The Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria for AUD of at least moderate severity (>3 symptoms)

Inclusion Criteria (Healthy Volunteer Participants):

1. Between the ages of 21 and 55
2. Right-handed
3. Able to perform informed consent and comply with study
4. Report drinking an average of fewer than 8/15 standard drinks per week for women/men and no more than 1 HDD (heavy drinking days) during the previous 28 days.

Exclusion Criteria (Participants with Alcohol use Disorder):

1. Neurological, medical or other conditions that would interfere with MRI scanning (e.g., history of stroke, seizure, brain tumor, brain infection, traumatic brain injury, multiple sclerosis, dementia, non MRI-compliant metal device in body, pregnancy, claustrophobia, color blindness, severe hearing impairment, weight>300 lbs., wheelchair-bound, tattoos as indicated by the guidelines established by the Zuckerman Institute MRI unit: https://mr.research.columbia.edu/
2. DSM 5 diagnoses of schizophrenia, schizoaffective disorder, or bipolar disorder
3. Any non-AUD psychiatric disorder that may, according to the investigator's judgment, require treatment over the course of the study
4. Significant suicide or violence risk
5. Currently taking psychotropic medication
6. Current substance use disorder other than AUD, tobacco use disorder or mild cannabis use disorder
7. Currently pregnant, attempting to become pregnant or nursing
8. Sufficiently socially unstable as to preclude participation (e.g. homeless).
9. Known history of allergy, intolerance, or hypersensitivity to disulfiram or its derivates
10. Contraindications to disulfiram treatment (e.g. liver disease, kidney disease, cardiac disease, seizure disorder, hypothyroidism, diabetes mellitus, pregnancy or lactation, allergy to disulfiram or thiuram derivatives)
11. Currently taking medications containing alcohol, metronidazole, isoniazid, paraldehyde, phenytoin, warfarin, or theophylline.
12. Treatment with concomitant medications that might interfere with disulfiram
13. A history of alcohol withdrawal seizures, delirium tremens or resistant alcohol withdrawal
14. Current moderate or severe alcohol withdrawal (CIWA >9 with BAL<0.05)
15. History of prior disulfiram treatment failure
16. Being abstinent for > 7 days at the time of screening

Exclusion Criteria (Healthy Volunteer Participants):

1. Neurological, medical or other conditions that would interfere with MRI scanning (e.g., history of stroke, seizure, brain tumor, brain infection, traumatic brain injury, multiple sclerosis, dementia, non MRI-compliant metal device in body, pregnancy, claustrophobia, color blindness, severe hearing impairment, weight>300 lbs., wheelchair- bound, tattoos as indicated by the guidelines established by the ZI MRI unit: https://mr.research.columbia.edu/
2. DSM 5 diagnoses of schizophrenia, schizoaffective disorder, or bipolar disorder
3. Any psychiatric disorder that may, according to the investigator's judgment, require treatment over the course of the study
4. Significant suicide or violence risk
5. Currently taking psychotropic medication
6. Current substance use disorder other than tobacco use disorder or mild cannabis use disorder
7. Currently pregnant, attempting to become pregnant or nursing
8. Sufficiently socially unstable as to preclude participation (e.g., homeless).
9. A diagnosis of AUD of any severity

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2029-08-30 (Estimated); Study Completion 2029-08-30 (Estimated)

PRIMARY OUTCOMES:
AI-BNST Resting state functional connectivity correlation (R) value | 1 week and 3 months
  Resting state functional connectivity between the bed nucleus of the stria terminalis and anterior insula resting state functional connectivity. Correlation values range from -1 to +1, with higher values indicating stronger connectivity.
AI-BNST task activation t statistic | 1 week and 3 months
  Unpredictable threat task activation of the bed nucleus of the stria terminalis and anterior insula. T statistics range from negative infinity to positive infinity. The farther the t statistic is away from zero (positively), this indicates a larger magnitude in brain activation
State trait anxiety inventory score | 1 week and 3 months
  The State-Trait Anxiety Inventory (STAI) score ranges from 20-80, with higher scores indicating greater anxiety

CONTACTS AND LOCATIONS:
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
fMRI data and metadata will be archived in OpenNeuro, and Electrodermal Activity data will be stored in the DANDI archive and deposited to NIAAA Data Archive (NIAAADA), which is part of the NIMH NDA. All data will be de-identified prior to receipt by the repository, but the information needed to generate a global unique identifier for the NIAAADA, which is part of the NIMH NDA, will be collected for each subject. Sufficient data from this project will be preserved to enable sharing via NIAAADA data of sufficient quality to validate and replicate research findings. NIAAA requires data measured from human subjects to be shared using the NIAAADA. All fMRI resting state and task related paradigm designs and experiment definitions will be deposited in the NIAAADA. Studies will be created that contain the data used for every publication. Sufficient data from this project will be preserved to enable sharing via NDA data of sufficient quality to validate and replicate research findings.
Time Frame: Data will be desposited after 12 months, uploaded every 6 months thereafter. The research community will have access to data. NIAAADA/NDA will make decisions about how long to preserve the data, but that data archive has not deleted any deposited data up to now.
Access Criteria: To request access of the data, researchers will use the standard processes at NIAAADA/NDA, and the NIAAADA/NDA Data Access Committee will decide which requests to grant. fMRI data will be publically available in OpenNeuro

REFERENCES:
- [Background] Anker JJ, Kushner MG, Thuras P, Menk J, Unruh AS. Drinking to cope with negative emotions moderates alcohol use disorder treatment response in patients with co-occurring anxiety disorder. Drug Alcohol Depend. 2016 Feb 1;159:93-100. doi: 10.1016/j.drugalcdep.2015.11.031. Epub 2015 Dec 11. PMID 26718394
- [Background] Anker JJ, Kushner MG. Co-Occurring Alcohol Use Disorder and Anxiety: Bridging Psychiatric, Psychological, and Neurobiological Perspectives. Alcohol Res. 2019 Dec 30;40(1):arcr.v40.1.03. doi: 10.35946/arcr.v40.1.03. eCollection 2019. PMID 31886106
- [Background] Glasser MF, Coalson TS, Robinson EC, Hacker CD, Harwell J, Yacoub E, Ugurbil K, Andersson J, Beckmann CF, Jenkinson M, Smith SM, Van Essen DC. A multi-modal parcellation of human cerebral cortex. Nature. 2016 Aug 11;536(7615):171-178. doi: 10.1038/nature18933. Epub 2016 Jul 20. PMID 27437579
- [Background] Brown SA, Irwin M, Schuckit MA. Changes in anxiety among abstinent male alcoholics. J Stud Alcohol. 1991 Jan;52(1):55-61. doi: 10.15288/jsa.1991.52.55. PMID 1994124
- [Background] Centanni SW, Morris BD, Luchsinger JR, Bedse G, Fetterly TL, Patel S, Winder DG. Endocannabinoid control of the insular-bed nucleus of the stria terminalis circuit regulates negative affective behavior associated with alcohol abstinence. Neuropsychopharmacology. 2019 Feb;44(3):526-537. doi: 10.1038/s41386-018-0257-8. Epub 2018 Nov 2. PMID 30390064
- [Background] Clauss JA, Avery SN, Benningfield MM, Blackford JU. Social anxiety is associated with BNST response to unpredictability. Depress Anxiety. 2019 Aug;36(8):666-675. doi: 10.1002/da.22891. Epub 2019 Apr 6. PMID 30953446
- [Background] Agarwal R, Sharma SK, Malaviya AN. Gold-induced hypersensitivity pneumonitis in a patient with rheumatoid arthritis. Clin Exp Rheumatol. 1989 Jan-Feb;7(1):89-90. PMID 2706825
- [Background] Driessen M, Meier S, Hill A, Wetterling T, Lange W, Junghanns K. The course of anxiety, depression and drinking behaviours after completed detoxification in alcoholics with and without comorbid anxiety and depressive disorders. Alcohol Alcohol. 2001 May-Jun;36(3):249-55. doi: 10.1093/alcalc/36.3.249. PMID 11373263
- [Background] Farb NA, Segal ZV, Anderson AK. Attentional modulation of primary interoceptive and exteroceptive cortices. Cereb Cortex. 2013 Jan;23(1):114-26. doi: 10.1093/cercor/bhr385. Epub 2012 Jan 19. PMID 22267308
- [Background] Flook EA, Feola B, Avery SN, Winder DG, Woodward ND, Heckers S, Blackford JU. BNST-insula structural connectivity in humans. Neuroimage. 2020 Apr 15;210:116555. doi: 10.1016/j.neuroimage.2020.116555. Epub 2020 Jan 16. PMID 31954845
- [Background] Joutsa J, Moussawi K, Siddiqi SH, Abdolahi A, Drew W, Cohen AL, Ross TJ, Deshpande HU, Wang HZ, Bruss J, Stein EA, Volkow ND, Grafman JH, van Wijngaarden E, Boes AD, Fox MD. Brain lesions disrupting addiction map to a common human brain circuit. Nat Med. 2022 Jun;28(6):1249-1255. doi: 10.1038/s41591-022-01834-y. Epub 2022 Jun 13. PMID 35697842
- [Background] Kushner MG, Abrams K, Thuras P, Hanson KL, Brekke M, Sletten S. Follow-up study of anxiety disorder and alcohol dependence in comorbid alcoholism treatment patients. Alcohol Clin Exp Res. 2005 Aug;29(8):1432-43. doi: 10.1097/01.alc.0000175072.17623.f8. PMID 16131851
- [Background] Schuckit MA, Hesselbrock V. Alcohol dependence and anxiety disorders: what is the relationship? Am J Psychiatry. 1994 Dec;151(12):1723-34. doi: 10.1176/ajp.151.12.1723. PMID 7977877
- [Background] Schuckit MA, Irwin M, Brown SA. The history of anxiety symptoms among 171 primary alcoholics. J Stud Alcohol. 1990 Jan;51(1):34-41. doi: 10.15288/jsa.1990.51.34. PMID 2299847
- [Background] Skinner MD, Lahmek P, Pham H, Aubin HJ. Disulfiram efficacy in the treatment of alcohol dependence: a meta-analysis. PLoS One. 2014 Feb 10;9(2):e87366. doi: 10.1371/journal.pone.0087366. eCollection 2014. PMID 24520330
- [Background] Srivastava AB, Sanchez-Pena J, Levin FR, Mariani JJ, Patel GH, Naqvi NH. Drinking reduction during cognitive behavioral therapy for alcohol use disorder is associated with a reduction in anterior insula-bed nucleus of the stria terminalis resting-state functional connectivity. Alcohol Clin Exp Res. 2021 Aug;45(8):1596-1606. doi: 10.1111/acer.14661. Epub 2021 Aug 2. PMID 34342012
- [Background] Theiss JD, Ridgewell C, McHugo M, Heckers S, Blackford JU. Manual segmentation of the human bed nucleus of the stria terminalis using 3T MRI. Neuroimage. 2017 Feb 1;146:288-292. doi: 10.1016/j.neuroimage.2016.11.047. Epub 2016 Nov 19. PMID 27876653
- [Background] Wilcox CE, Dekonenko CJ, Mayer AR, Bogenschutz MP, Turner JA. Cognitive control in alcohol use disorder: deficits and clinical relevance. Rev Neurosci. 2014;25(1):1-24. doi: 10.1515/revneuro-2013-0054. PMID 24361772